CLINICAL TRIAL: NCT04856709
Title: Abdominal Pectopexy Versus Abdominal Sacral Hysteropexy as Conservative Surgeries for Genital Prolapse: A Randomized Control Trial
Brief Title: Abdominal Pectopexy Versus Abdominal Sacral Hysteropexy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pectopexy
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Genital Prolapse

STUDY DESIGN:
Intervention Model Description: * Study design: Randomized Controlled clinical Trial
  * Study Setting: Ain Shams maternity hospital.
  * Study Population: The study included 80 women divided into 2 groups:
  Group A: 40 women underwent abdominal pectopexy. Group B: 40 women underwent abdominal sacral hysteropexy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): Women with stage 2 to 4 uterine prolapse. BMI from ≤ 35 kg\m2. Women of any parity including nulliparas will be included. Age of female patients ranges from 20 to 40 years.
  Interventions: Procedure: Abdominal Pectopexy; Procedure: Abdominal Sacral Hysteropexy

INTERVENTIONS:
Procedure: Abdominal Pectopexy — Pectopexy is a new technique for apical repair in which lateral parts of the iliopectineal ligament are used for cuff or cervix suspension.
Procedure: Abdominal Sacral Hysteropexy — Abdominal sacrocolpopexy is a procedure that uses a mesh material to support the top of the vagina to treat pelvic prolapse.

SUMMARY:
This study aims to compare between abdominal pectopexy and abdominal sacral hysteropexy in terms of efficacy (assessed by POP-Q system), intra and postoperative complications.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP), the herniation of the pelvic organs to or beyond the vaginal walls, is a common condition. Many women with prolapse experience symptoms that impact daily activities, sexual function, and exercise. The presence of POP can have a detrimental impact on body image and sexuality (Lowder et al., 2011). Nulliparous prolapse is reported to account for 1.5% to 2% of all cases of genital prolapse (Virkud, 2016). The incidence rises to 5 -8 % for young women who have delivered one or two children. As this type of prolapse occurs at a younger age, the surgical technique should not only reduce the prolapse but also retain the reproductive function. Various conservative surgeries have been described in the past, each having their own merits and de-merits (Rameshkumar et al., 2017).

Pelvic organ prolapse (POP) is affecting women of all ages. Epidemiological studies suggest a lifetime risk of prolapse or incontinence surgery of between 7 and 19% (Olsen et al., 1997; Smith et al., 2010). In an ageing population, the incidence of these surgeries would only be expected to increase, although the increasing Caesarean Section rates and smaller family size in recent years will have a negative impact on the prevalence of these conditions. There are many approaches to the surgical correction of POP, which frequently reflect the nature and anatomical site of the defective support, but essentially the surgeon has to decide whether to perform this surgery vaginally or via the abdomen as an open or laparoscopic procedure. If performed vaginally, further decisions regarding the use of synthetic or biological graft to reinforce the repair need to be made (Cvach and Dwyer, 2012).

Pectopexy is a new technique for apical repair in which lateral parts of the iliopectineal ligament are used for cuff or cervix suspension. This new method is considered a simple, safe procedure, especially in patients whose surgical exploration is difficult (Banerjee and Noé, 2011).

This method uses the iliopectineal ligament on both sides for the mesh ﬁxation, (Banerjee and Noé, 2011). so there is no restriction caused by the mesh. The mesh follows natural structures (round and broad ligaments) without crossing sensitive spots, such as the ureter or bowel. The hypogastric trunk is at a safe distance and out of danger.

The iliopectineal ligament is an extension of the lacunar ligament that runs on the pectineal line of the pubic bone (Faure et al., 2001), and is significantly stronger than the sacrospinous ligament and the arcus tendineus of the pelvic fascia (Cosson et al., 2003). The structure is strong, and holds suture well Abdominal sacral hysteropexy remains a viable alternative for women undergoing pelvic reconstructive surgery who wish to retain their uteri, providing comparable rates of overall improvement and symptom change. Avoiding hysterectomy decreases the risk of mesh erosion but may increase the risk of subsequent recurrent prolapse, specifically in the anterior compartment (Cvach and Cundiff, 2008).

Although sacrocolpopexy has been the most effective option over time, the procedure is still associated with some problems, and the most frequently reported complications include defecation disorders and stress urinary incontinence (SUI)

ELIGIBILITY:
Inclusion Criteria:

* Women with stage 2 to 4 uterine prolapse.
* BMI from ≤ 35 kg\m2.
* Women of any parity including nulliparas will be included.
* Age of female patients ranges from 20 to 40 years.

Exclusion Criteria:

* Previous correction of apical prolapse.
* Inoperable co-existing uterine pathology

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Efficacy, After the procedure there will be follow up visits at 3 months to detect the efficacy of the procedure by using POP-Q system. | 3 months
  The POP-Q system is a technique that measures compartment prolapse relative to the anatomic landmark of the hymen.Prolapse points proximal to the hymen are given a negative value, whereas positive values are given to points that protrude past the hymen. 6 points are delineated, including two on the anterior vaginal wall (Aa, Ba), two on the vaginal apex (C, D), and two on the posterior vaginal wall (Ap, Bp). Points Gh, Pb, and TVL describe the genital hiatus, perineal body, and total vaginal length, respectively.
  * Stage 0: no demonstrable prolapse
  * Stage 1: the most distal portion of the prolapsed segment is >1 cm above the level of the hymen
  * Stage 2: the most distal portion of the prolapsed segment is >1 cm or less proximal or distal to the hymen
  * Stage 3: the most distal portion of the prolapsed segment protrudes >1 cm below the hymen but 2 cm less than the total length of the vagina
  * Stage 4: complete eversion of the vagina

SECONDARY OUTCOMES:
Operative time | 60- 240 minutes
  Total operative time from skin incision till closure of the skin and excluding time of concomitant surgical procedures.
Intra operative blood loss | 60- 240 minutes
  Intra operative blood loss will be estimated via:
  Amount of blood in suction bottle. Drop in postoperative hemoglobin and hematocrit when compared with preoperative values
Intra operative complications | 60- 240 minutes
  Intra operative complications including:
  * Need for blood transfusion.
  * Bowel or bladder injury.
Post operative complications | 1 week
  * Subfascial hematoma or pelvic hematoma.
  * Surgical site infection.
  * Urinary tract infection.
  * Need for post-operative blood transfusion.
  * Postoperative bowel or urinary tract complications
Post operative pain | after 6 hours, 12 hours and 24 hours from the operation
  Postoperative pain will be assessed using the linear 10cm visual analogue scale. Range is from 10(unbearable pain) to zero (no pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication